CLINICAL TRIAL: NCT05729178
Title: Unravelling the Role of KCTD Protein Family in the Clinical Management of Childhood Acute Lymphoblastic Leukemias
Status: Recruiting | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Collaborators: Santobono-Pausilipon Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 5/19
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-02

CONDITIONS: Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric acute lymphoblastic leukemia patients: pediatric patients of 1-16 years old affected by acute lymphoblastic leukemia
  Interventions: Other: observational study
- healthy subjects: cord blood from healthy donors that cannot be used for clinical purposes
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — analysis of biomarkers of interest (DNA-RNA and proteins) in MNC purified from the subjects' blood

SUMMARY:
A transcriptomic analysis of bone marrow from B-ALL patients was performed by our research group for identifying novel protein/factor with a putative role of disease biomarker. Along with some already known B-ALL biomarkers, our analysis highlighted deregulation of some members of an emerging protein class denoted as KCTD (Potassium ChannelTetramerization Domain-containing proteins). Starting from our preliminary observations, and considering that KCTDs havenever been studied in ALL, we decided to study these proteins in B- and T-ALL affected pediatric patients, enrolled by our research group in collaboration with AORN Santobono-Pausilipon pediatric oncological hospital.Indeed, the present research program aims at opening a new scenario for the study of KCTD proteins in childhood leukemias. The final goal of the project will be to evaluate the translational relevance of selected deregulated KCTDs as novel biomarkers useful for B-ALL and T-ALL diagnostics, and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-18 years of both sexes diagnosed with B- ALL and T-ALL;
* Patients who will have signed the informed consent

Exclusion Criteria:

* Patients who refuse to participate in the study;
* Patients who do not fall within the age range mentioned above

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study foresees the possibility of recruiting approximately 60 patients with B-ALL and 15-20 patients with T-ALL. Furthermore, control subjects with age and sex comparable to those of the patients will be recruited. Finally, about 100 units of cord blood that do not meet the criteria for therapeutic cryopreservation and for which consent has been given for their use for scientific research will be used
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
KCTD expression levels, by RNAseq approach, in a cohort of B and T cell ALL affected patients compared to unaffected controls | 1-12 months
  We enroll during this project about 15-20 B-ALL, and 3-6 T-ALL patients.RNAseq experiments for transcriptome analysis will be performed on a study cohort of at least 8 B-ALL patients, 3-4 T-ALL patients, and naive B or T cells purified from cord blood as control for B- and T-ALL correspondingly. Raw counts will be used and an empirical Bayes approach applied (DESeq2, R package). The results will include, for each gene, log-fold change (log2), base mean, p-value and adjusted p-values (Benjamimi-Hochberg). DEgenes output will be exported into format suitable for IPA Ingenuity pathway AnalysisSoftware (Qiagen), for gene annotations, functional analysis and biomarker prediction. The KCTD proteins that will be dereguleted in B-ALL and T-ALL will be studied in detail.
RT-PCR validation of deregulated KCTDs and identification of possible KCTDs interactors in leukemia by functional proteomic approach | 13-24 months
  After the interpretation of transcriptome data we will perform specific validation experiments by reat-time pcr, westernblotting, flow cytometry and microscopy. Briefly,total RNA will be purified from about 5e6 total MNC and used for RT-PCR experiments; BM smear will be collected for immunofluorescence analysis of deregulated KCTDs; protein total extract will be obtained from at least 1 e 6 total MNC and stored at -80°C until Western Blotting; finally, live mononuclear cells will be treted for permeabilization and cytoplasmic immunostaining of the KCTDs of interest. All experiments will be settled-up on B- and T-ALL in vitro human model systems and then performed on patients and controls cells. Moreover, in order to identify possible interactors of KCTDs proteins we will use B-ALL and T-ALL cell lines for functional proteomics analysis.
Correlation of B-ALL patients clinical data with KCTDs expression level | 25-36 months
  Firstly, we will evaluated the usefulness of the deregulated KCTD proteins as novel markers of leukemia to be tested by multiparametric clinical flowcytometry. A specific protocol has been already setted-up by our research team, and it is able to stain cytoplasmicantigens (such as KCTD proteins) with surface antigens commonly used for to study hematoogical compartments by flowcytometry. This approach will be useful especially in monitoring patient response to treatment as well as detection of minimal residual disease. Moreover, being able to detect cytoplasmic KCTDs in combination with surface antigens, we planned to describe the KCTDs expression levels in multiple cellular population residing in marrow and peripheral blood.Secondly, the overall data obtained in this study will be also interpreted looking at the patient clinics with particular reference to the response to therapy, the risk of relapse and, when possible, resistance to therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Synlab SDN, Naples, Italy

IPD SHARING:
Plan to Share IPD: No